CLINICAL TRIAL: NCT01841008
Title: Maintenance Treatment of Non Segmental Vitiligo With Tacrolimus Ointment 0.1% Versus Control, Randomized and Double Blind Study
Brief Title: Maintenance Treatment of Non Segmental Vitiligo With Tacrolimus Ointment 0.1% Versus Control
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-PP-12
Record Dates: First submitted 2012-03-23; First posted 2013-04-26 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-06

CONDITIONS: Pigmentation Disorders; Vitiligo
Keywords: [C17.800.621]
MeSH Terms: conditions — Pigmentation Disorders; Vitiligo | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus ointment 0.1% (Experimental)
  Interventions: Drug: Protopic
- Group Placebo (Placebo Comparator)
  Interventions: Drug: Placebo : Diprobase

INTERVENTIONS:
Drug: Protopic — Topical treatment (tacrolimus or placebo) will be delivered to the patient by the hospital pharmacy and should be applied twice per week (3 or 4 days apart) for 24 weeks.
  Arms: Tacrolimus ointment 0.1%
Drug: Placebo : Diprobase — Topical treatment (tacrolimus or placebo) will be delivered to the patient by the hospital pharmacy and should be applied twice per week (3 or 4 days apart) for 24 weeks.
  Arms: Group Placebo

SUMMARY:
Tacrolimus ointment 0.1% has shown promising results for treating vitiligo in many prospective studies. Prospective randomized studies versus placebo are required to confirm the hypothesis that maintenance treatment with two applications of tacrolimus ointment 0.1% per week can reduce relapses of non-segmental vitiligo lesions.

Main objective To assess the efficacy of maintenance therapy with topical tacrolimus vs placebo in the prevention of depigmentation in patients with vitiligo who responded to treatment.

Secondary objectives

* Evaluate the efficacy of maintenance therapy with tacrolimus vs topical placebo to decrease the intensity of depigmentation in patients with vitiligo who responded to treatment.
* To study the occurrence of possible adverse effects.

Length of the study Inclusion: 12 months Treatment: 6 months Follow-up: 6 months Total length of the study: 18 months

Intervention Multicentric prospective interventional randomized comparative study versus placebo.

* Visit V0: Selection Information of the patient, control of inclusion and non inclusion criteria.
* Visit V1: Control of inclusion and non inclusion criteria, patients signed informed consent. An initial clinical evaluation and photographs in direct sunlight and UV. Topical treatment (tacrolimus or placebo) will be delivered to the patient by the hospital pharmacy and should be applied twice per week (3 or 4 days apart) for 24 weeks.
* Visit V2:

The patient will be reviewed after the end of treatment (24 weeks after the visit V1) for final evaluation. A clinical assessment will be made and photographs in the same way as the inclusion. Adverse reactions during treatment will be collected by the investigator (they will be noted as and when the patient in a notebook that will be presented at baseline).

The percentage of depigmentation will be evaluated in a blinded treatment of photographs by two reviewers. In case of disagreement, the opinion of a third appraiser will be required.

- End of study: After the end of the study patients will be supported via the usual care recommended for their condition.

Evaluation criteria

* primary endpoint

  ---Percentage of patients at 24 weeks without depigmentation (depigmentation score = 0). A score of depigmentation from 0 to 2 will be used. A blind treatment evaluation of direct light and UV photographs will be made by two independent observers (dermatologists) between inclusion and after 24 weeks of treatment.
* secondary endpoints

  ---- The efficiency to reduce the intensity of relapses will be evaluated using the score of depigmentation (rate of patients with a score of 0 or 1 in each group) and the VASI score (Appendix 4).
* The frequency, severity and time of occurrence of adverse events are reported. Side effects are classified into grades according to WHO criteria.

Number of subject Considering that depigmentation occurs in more than 40% of patients during the 24 weeks of maintenance treatment and hoped that the proactive treatment will reduce the rate of depigmentation of 10%, a population of 26 patients per group will be necessary (taking into account 10% of patients lost to follow). The total number of patients to be included in the study will be 52.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Non-segmental vitiligo repigmented more than 75% with treatment (any type of treatment is accepted: NB-UVB, PUVA, lamp or excimer laser at 308 nm, topical steroids, topical tacrolimus, graft). The total area treated plates during maintenance treatment should not exceed 10% of the total body surface area.
* Affiliation to the Social Security
* Informed consent signed by the patient

Exclusion Criteria:

* Segmental Vitiligo
* Pregnant or breastfeeding women (pregnancy test will be conducted); effective contraception will be maintained for the duration of the study.
* Allergy to macrolide derivatives.
* Exposure to UV or concomitant exposure to the sun without protective shield.
* Concomitant immunosuppressive therapy or oral corticosteroids for topical (on the vitiligo lesions) or systemic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
UV and direct light photographs | At 6 months
  Comparison of photographs between day 0 and 24 weeks by two independent-blinded dermatologists

SECONDARY OUTCOMES:
Score of depigmentation, VASI score. Frequency and severity of adverse events. | At 6 months
  Score of depigmentation, VASI score. Frequency and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, Pu-Ph, Principal Investigator — CHU de Nice - Service de Dermatologie - Hôpital de l'Archet - 151 Route de saint-antoine de ginestière 06200 Nice
Locations (2):
- France (2):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes
  - CHU de Bordeaux, Bordeaux, Gironde